CLINICAL TRIAL: NCT06229457
Title: Development and Feasibility Testing of a Boys & Girls Clubs' Sports Intervention to Promote Physical Activity in Rural Girls: Girls PLAY
Brief Title: Development and Testing of a Sports Intervention to Promote Physical Activity in Rural Girls
Acronym: GirlsPLAY
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Boys and Girls Clubs of Imperial Valley (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS-2023-0186; 1K01HL171860-01 (NIH)
Record Dates: First submitted 2024-01-11; First posted 2024-01-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Girls PLAY program (Experimental)
  Interventions: Behavioral: Girls PLAY program

INTERVENTIONS:
Behavioral: Girls PLAY program — Girls PLAY program (8-12 weeks) will include 1) a series of in-person sessions, led by Boys and Girls Clubs staff at the Boys and Girls Club sites, and 2) take-home activities. In-person sessions (60-75 min; 2-3x/week) will center around a different developmentally appropriate sport each week. Lesson plans will outline games/activities in which youth engage in fundamental, sport-specific movement skills. Lesson plans will be delivered by Boys and Girls Club leaders using acts of instruction derived from Self-Determination Theory. Take home activities will 1) summarize and add on to the week's in-person sessions and 2) be adapted for delivery by parents and/or self-guided participation by youth. Take-home activities will provide information for engaging in the past week's activities as well as additional activities that parents and youth can participate in together.

SUMMARY:
The goal of this study is to examine the impact of a 12-week sports sampling and physical literacy program on rural girls' physical activity.

DETAILED DESCRIPTION:
Fewer than 30% of elementary-aged youth meet physical activity guidelines, with lower activity levels found among girls, racial minorities, and those living in rural areas. Sport is one of the best strategies for promoting physical activity, yet girls, Hispanics, and rural populations participate in youth sport at lower numbers and drop out at a higher rate. In line with Self-Determination Theory, commonly cited barriers include lack of competence, autonomy, and relatedness. Physical literacy and sport sampling have also been identified as key determinants of youth sport participation. Developing interventions around physical literacy and sport sampling, with intervention delivery grounded in Self-Determination Theory principles, is a promising strategy for promoting youth sport. However, the few existing interventions aimed to promote girls' physical activity through sport were developed outside the United States, focused on adolescent (versus younger) girls, and/or conducted among urban or suburban youth, limiting generalizability. Rural, Hispanic girls face unique challenges around sport that should be identified and addressed, yet there remains a paucity of information on determinants of sport participation among this population.

This study aims to to develop, tailor, and examine the impact of a tailored Boys & Girls Clubs (BGC) sport sampling and physical literacy program on rural girls' physical activity levels. BGC is an organization that provides learning and leadership programs to millions of rural youth nationwide, about half of whom are girls.

This study will enroll Hispanic girls ages 8-10 living in rural Imperial County, California. The first aims are to develop and refine a 12-week sport sampling and physical literacy intervention entitled "Girls Positive Learning Activities for Youth", or "Girls PLAY". The Girls PLAY intervention will be delivered as Boys & Girls Clubs programming, and intervention delivery will be grounded in Self-Determination Theory. We will then examine the feasibility of the 12-week Girls PLAY intervention. Secondary outcomes of physical activity levels, physical literacy, Self-Determination Theory constructs, and sports participation will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* living in Imperial County, California
* identify as female
* aged 8-10 years old
* enrolled at a participating Boys & Girls Club site

Exclusion Criteria:

* has a sibling enrolled in the study
* physical or mental impairment that would preclude physical activity or protocol compliance

Ages: 8 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Recruitment capability | Weeks 10-12
  Feasibility metric: successfully enroll 30 participants
Study assessments completed | Weeks 10-12
  Feasibility metric: ≥75% participants complete time 1 and time 2 assessments
Intervention acceptability and appropriateness | Weeks 10-12
  Feasibility metric: Mean score ≥3 on the Acceptability of Intervention Measure; mean score ≥3 on the Intervention Appropriateness Measure
Intervention feasibility and participant attendance | Weeks 10-12
  Feasibility metric: Mean score ≥3 on the Feasibility of Intervention Measure
Participant attendance | Weeks 10-12
  Attend ≥75% of in-person sessions (on average)

SECONDARY OUTCOMES:
Change from baseline in physical activity levels at 10-12 weeks measured via Actigraph GT3X+ | Week 0-1; Week 10-12
  We will use Actigraph GT3X+ (ActiGraph LLC, Pensacola, FL) to obtain a valid, objective measure of physical activity. Data will be collected over 7 days (sample frequency of 30 Hz; 15-sec epochs).
Change from baseline in physical literacy at 10-12 weeks measured via the Canadian Assessment for Physical Literacy, Second Edition (CAPL-2) | Week 0-1; Week 10-12
  Physical literacy changes will be assessed using the Canadian Assessment for Physical Literacy, Second Edition (CAPL-2). This includes the plank, Progressive Aerobic Cardiovascular Endurance Run, Canadian Agility & Movement Skill Assessment, and 22-item questionnaire.
Change from baseline in autonomy at 10-12 weeks | Week 0-1; Week 10-12
  Autonomy will be measured using the 9-item Autonomy-Supportive Coaching Questionnaire.
Change in sport engagement at 10-12 weeks | Week 0-1; Week 10-12
  Engagement will be assessed via child survey examining current sport involvement (length of involvement, primary and secondary sport) and behavioral intention (e.g., "I intend to play sports this year") adapted from items used in studies among similar age groups.
Change in sport enjoyment at 10-12 weeks | Week 0-1; Week 10-12
  Enjoyment will be assessed using an adapted 5-item Enjoyment subscale of the Sport Commitment Questionnaire-2.
Change from baseline in competence at 10-12 weeks | Week 0-1; Week 10-12
  Competence will be measured using an adapted version of the Perceived Competence Scale (4-item).
Change from baseline in relatedness at 10-12 weeks | Week 0-1; Week 10-12
  Relatedness will be measured using a 5-item acceptance subscale of the Need for Relatedness Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

REFERENCES:
- [Derived] Johnson A, Bocarro J, Kroshus-Havril E, Arredondo E. Development and testing of a sports intervention (Girls PLAY)to promote physical activity among rural girls: a feasibility study protocol. Pilot Feasibility Stud. 2026 Feb 2. doi: 10.1186/s40814-026-01765-2. Online ahead of print. PMID 41630110